CLINICAL TRIAL: NCT06665607
Title: Effects of Intrinsic Foot Muscles Training in Improving Stability in Multiple Sclerosis Patients
Brief Title: Foot Muscles Training in Sclerosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inés Llamas-Ramos (Other)
Responsible Party: Sponsor-Investigator, Inés Llamas-Ramos, PhD, University of Salamanca
Organization: University of Salamanca (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FOOT TRAINING-SCLEROSIS
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Multiple Sclerosis; Muscle Weakness; Training Group, Sensitivity
MeSH Terms: conditions — Multiple Sclerosis; Muscle Weakness; Hypersensitivity

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Training Group (Experimental)
  Interventions: Procedure: Intrinsic Mucle Training
- Control Group (Sham Comparator)
  Interventions: Procedure: Intrinsic Mucle Training

INTERVENTIONS:
Procedure: Intrinsic Mucle Training — Conventional physiotherapy treatment and the intrinisc foot muscles strengthening program for 8 weeks.

SUMMARY:
The study tries to assess the efficacy of an 8-week IFM training programme on stability in patients diagnosed with Multiple Sclerosis

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate neurological disability as scored by the Expanded Disability Status Scale (EDSS), ranging from 3.0 to 6.0

Exclusion Criteria:

* Cognitive disturbances that could affect the performance of any of the tests or questionnaires included in the study
* Diagnosis of visual or vestibular disorders that could affect patient stability
* Change in Multiple Sclerosis-specific medication in the 2 months prior to the start of the study
* Acute relapse in the 2 months prior to the start of the study
* Traumatologic or orthopaedic disorders that could negatively affect balance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-11-04 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Four Square Step Test (FSST): dynamic stability assessment test. | Initial and after 8 weeks
  The test consists of drawing a cross on the floor, delimiting 4 squares. The subject is placed in square number 1 in front of square number 2. The objective is to enter as quickly as possible into each square following the following sequence: Square number 1, 2, 3, 4, 1, 4, 4, 3, 2 and 1. It measures time.
Six Spot Step Test (SSST): test that quantitatively assesses lower limb function | Initial and after 8 weeks
  The test field measured one meter (width) by five meters (length). In the middle of the width line (0.50 m), a cone was placed in the proximal and distal areas of the line (start point and finish point). On each lateral line, two cones were placed at distances of one and three meters on the left. Another two cones were placed at two and four meters on the right. The subjects were instructed to walk on alternating sides and to kick the cones, alternating between the medial and lateral sides of the same foot. The subjects were instructed to complete the test as quickly as possible, without running. It measures distance.
The Frailty and Injuries: Cooperative Studies of Intervention Tecnhiques (FICSIT-4 test): Test of static balance | 0-9 points. Initial and after 8 weeks
  Participants have to maintain four progressively difficult foot positions for 10 seconds each (side by side stance, semi-tandem stance, tanden stance, unipedal stance). It measures the ability to maintain posture without losing balance is evaluated.
Activities-specific Balance Confidence scale (AsBC) | Initial and after 8 weeks
  Evaluate the patient´s perceived of balance confidence during 16 different daily activities. 0%-100%

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No